CLINICAL TRIAL: NCT00077675
Title: A Phase 2, Randomized, Double-Blind, Multinational Trial of Intravenous Telavancin Versus Standard Therapy for Treatment of Complicated Gram-Positive Skin and Skin Structure Infections (Gram Positive cSSSI)
Brief Title: Phase 2 Trial of TD-6424 (Telavancin) Versus Standard Therapy for Complicated Gram Positive Skin and Skin Structure Infections (Gram Positive cSSSI)
Acronym: FAST2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Steven Barriere, Pharm.D., Vice President, Clinical and Medical Affairs, Theravance, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: I6424-202b
Record Dates: First submitted 2004-02-10; First posted 2004-02-13 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Infections, Gram-positive Bacterial
Keywords: Abscess; Burns; Cellulitis; Ulcer; Wound infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Abscess; Burns; Cellulitis; Ulcer; Wound Infection | interventions — telavancin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telavancin (Experimental)
  Interventions: Drug: Telavancin
- Standard of care for cSSSI (Active Comparator): cSSSI - comlicated skin and skin structure infections
  Interventions: Drug: vancomycin or antistaphylococcal penicillin

INTERVENTIONS:
Drug: Telavancin — Telavancin 7.5 mg/kg/day, amended to 10 mg/kg/day, IV (intravenously) for up to 14 days
  Other Names: TD-6424; VIBATIV
  Arms: Telavancin
Drug: vancomycin or antistaphylococcal penicillin — Vancomycin 1 Gram IV (intravenously) every 12 hrs or nafcillin 2 Grams, oxacillin 2 Grams, or (in South Africa) cloxacillin 0.5 - 1 Gram, IV (intravenously) every 6 hrs for up to 14 days.
  Arms: Standard of care for cSSSI

SUMMARY:
Serious infections caused by resistant bacteria are becoming more of a medical problem throughout the world. This study will measure how well TD-6424 (Telavancin) can control infections and whether the drug is safe to give to patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of one of the following complicated skin and soft tissue infections and either a suspected or confirmed Gram positive organism

  * major abscess requiring surgical incision and drainage
  * infected burn (see exclusion criteria for important qualifications)
  * deep/extensive cellulitis
  * infected ulcer (see exclusion criteria for important qualifications)
  * wound infection
* Patients must be expected to require at least 4 days of intravenous (IV) antibiotic treatment

Exclusion Criteria:

* Previous systemic antibacterial therapy (with the exception of aztreonam and metronidazole) for > 24 hours within 7 days prior to the first dose of study drug unless the pathogen was resistant to prior treatment or the patient was a treatment failure (no clinical improvement after 3 days)
* Burns involving > 20% of body surface area or third degree/full thickness in nature, diabetic foot ulcers, ischemic ulcers/wounds, necrotizing fasciitis, gas gangrene, or mediastinitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2004-02; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Ralph Corey, MD, Principal Investigator — Duke University
Locations (1):
- Paradise Valley Hospital, 2400 E. 4th Street, National City, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: 20Feb2004 to 09SEP2004
Groups:
- Telavancin: Telavancin 10 mg/kg every 24 hours intravenously
- Standard of Care for cSSSI: Standard therapy [nafcillin or oxacillin 2 gram, or cloxacillin (in S. Africa) 0.5 to 1.0 gram, every 6 hours, or vancomycin 1 gram every 12 hours, intravenously]
Period: Overall Study
Arm/Group | Telavancin | Standard of Care for cSSSI
Started | 103 | 98
Completed | 92 | 89
Not Completed | 11 | 9
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 6 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 0 | 1
Not completed — Never received study treatment | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telavancin | Standard of Care for cSSSI | Total
Number analyzed (Participants) | 100 | 95 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92 | 91 | 183
  >=65 years | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (13.7) | 42.3 (10.8) | 43.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 33 | 78
  Male | 55 | 62 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 17 | 31
  Not Hispanic or Latino | 86 | 78 | 164
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 29 | 30 | 59
  White | 41 | 43 | 84
  More than one race | 24 | 19 | 43
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 54 | 112
  South Africa | 42 | 41 | 83
Diabetes Status [Number; unit: participants]
  Diabetic | 18 | 14 | 32
  Not Diabetic | 82 | 81 | 163

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Which is Measured at Test of Cure (TOC) in the Clinically Evaluable (CE) Population
Description: * Cure: Resolution of clinically significant signs, symptoms associated with the skin infection present at study admission or improvement to the extent that the infectious process had been controlled and no further therapy with study medication was necessary.
  * Failure: Inadequate response to study therapy or the need for significant surgical management (e.g. more than just routine debridement) of the infection site following antibiotic therapy and prior to Test-of-Cure (TOC) visit
  * Indeterminate: Inability to determine outcome.
Time Frame: 7 to 14 days following completion of antibiotic treatment
Population: The CE population was a subset of the All Treated Population and was composed of patients who met the inclusion/exclusion criteria or were granted permission to enroll and had a clinical response of "cure" or "failure." The All Treated Population patients received at least one treatment. The Primary Efficacy Analysis was of the CE population.
Measure: Number; unit: participants
Arm/Group | Telavancin | Standard of Care for cSSSI
Number analyzed (Participants) | 77 | 77
participants
  Cured | 74 | 72
  Failure | 3 | 5
Statistical Analysis 1: Comparison: Telavancin vs Standard of Care for cSSSI; 95% Confidence Interval: -0.0527 to 0.1102 No estimated value Parameter that was estimated: Risk Difference; Test type: Non-Inferiority or Equivalence — Sample size was selected on the basis of clinical judgment and was deemed adequate to provide clinically meaningful descriptive results consistent with study objectives. This sample size was estimated to provide 91% power to test telavancin's non-inferiority to vancomycin with respect to clinical response using a non-inferiority margin of 20%; p = 0.5318, 2-sided 95% confidence interval calculat

ADVERSE EVENTS:
Description: The Safety Population was the "All Treated Population" - all patients who received one treatment. The Primary Analysis was of the Clinically Evaluable (CE) Population. The CE population was composed of the patients who met the inclusion / exclusion criteria or were granted permission to enroll and had a clinical response of "cure" or "failure".
Arm/Group | Telavancin | Standard of Care for cSSSI
Serious Adverse Events (participants affected / at risk) | 7/100 | 3/95
Other Adverse Events (participants affected / at risk) | 56/100 | 54/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=100) | Standard of Care for cSSSI (N=95)
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Ileostomy (Surgical and medical procedures) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Wound Haemorrhage (Vascular disorders) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Multi-organ Failure (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=100) | Standard of Care for cSSSI (N=95)
Anemia (Blood and lymphatic system disorders) | 3 | 4
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Eye Irritation (Eye disorders) | 1 | 0
Eye Swelling (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 5 | 7
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 16 | 6
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 6
Application Site Erythema (General disorders) | 0 | 1
Application Site Pruritus (General disorders) | 0 | 1
Catheter Site Inflammation (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 2
Chills (General disorders) | 6 | 2
Drug Withdrawal Syndrome (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Infusion site bruising (General disorders) | 1 | 0
Infusion site burning (General disorders) | 2 | 1
Infusion site erythema (General disorders) | 1 | 3
Infusion site induration (General disorders) | 1 | 0
Infusion site pain (General disorders) | 1 | 0
Infusion site phlebitis (General disorders) | 1 | 0
Infusion site rash (General disorders) | 0 | 1
Infusion site swelling (General disorders) | 1 | 0
Multi-organ Failure (General disorders) | 0 | 1
Night sweats (General disorders) | 2 | 0
Oedema Peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 4
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0
Central Line Infection (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 0
Fungal Infection (Infections and infestations) | 1 | 2
Fungal skin infection (Infections and infestations) | 1 | 0
Herpes Simplex (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
HIV Infection (Infections and infestations) | 3 | 0
Infection (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 1 | 0
Oral Candidiasis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 1
Tinea Infection (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 2
Urinary Tract Infection Fungal (Infections and infestations) | 1 | 0
Vaginal mycosis (Infections and infestations) | 1 | 1
Wound Infection (Infections and infestations) | 1 | 2
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0
Activated Partial Thromboplastin Time (Investigations) | 0 | 1
Alanine Aminotransferase increased (Investigations) | 3 | 1
Albumin Urine Present (Investigations) | 3 | 0
Aspartate Aminotransferase increased (Investigations) | 3 | 1
Bacteria Urine (Investigations) | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 3
Blood Bilirubin Increased (Investigations) | 0 | 1
Blood Creatinine Increased (Investigations) | 3 | 1
Blood Glucose increased (Investigations) | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 3
Blood Magnesium decreased (Investigations) | 1 | 0
Blood Urea increased (Investigations) | 1 | 0
Eosinophil Count increased (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 5
Hepatic Enzyme increased (Investigations) | 0 | 9
Liver function test abnormal (Investigations) | 0 | 2
Nitrite Urine present (Investigations) | 0 | 1
Platelet count increased (Investigations) | 2 | 0
Prothrombin time prolonged (Investigations) | 1 | 1
QRS axis abnormal (Investigations) | 0 | 1
Respiratory rate increased (Investigations) | 1 | 0
Urinary casts (Investigations) | 2 | 0
Urine analysis abnormal (Investigations) | 3 | 0
White Blood Cell Count decreased (Investigations) | 0 | 1
White Blood Cell Count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 6
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Ageusia (Nervous system disorders) | 1 | 0
Depressed Level of Consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 2
Dizziness Postural (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 14 | 0
Headache (Nervous system disorders) | 8 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 1
Paraesthesia oral (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Affect Lability (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 13 | 3
Suicidal Ideation (Psychiatric disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 4 | 2
Microalbuminuria (Renal and urinary disorders) | 3 | 5
Pyuria (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Genital Burning Sensation (Reproductive system and breast disorders) | 1 | 0
Genital Pruritis Female (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Crackles Lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 6 | 8
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Ileostomy (Surgical and medical procedures) | 1 | 0
Intubation (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Hot Flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 1
Hypotension (Vascular disorders) | 2 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 2
Wound Haemorrhage (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less